CLINICAL TRIAL: NCT01810380
Title: Interventional, Randomised, Double-blind, Parallel-group, Placebo-controlled, Active-reference, Flexible-dose Study of Brexpiprazole in Patients With Acute Schizophrenia
Brief Title: Brexpiprazole in Patients With Acute Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14644A; 2012-002252-17 (EudraCT Number)
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Brexpiprazole (Experimental): Patients randomised to brexpiprazole received 1mg/day on Day 1, 2mg/day on Day 2, 3mg/day on Day 3 (uptitration); the dose could be adjusted from Day 4 onwards to 2, 3, or 4mg/day to optimise the clinical effect and tolerability.
  Interventions: Drug: Brexpiprazole
- Quetiapine extended release (Other): Active Reference. Patients randomised to quetiapine received 300mg/day on Day 1, 600mg/day on Days 2 and 3 (uptitration); the dose could be adjusted from Day 4 onwards to 400, 600, or 800mg/day to optimise the clinical effect and tolerability.
  Interventions: Drug: Quetiapine extended release

INTERVENTIONS:
Drug: Placebo — Once daily as tablets and capsules, orally
  Arms: Placebo
Drug: Brexpiprazole — 2-4 mg/day, once daily, tablets, orally
  Arms: Brexpiprazole
Drug: Quetiapine extended release — 400-800 mg/day, once daily, encapsulated tablets, orally
  Other Names: Seroquel XL®/XR®
  Arms: Quetiapine extended release

SUMMARY:
To determine the efficacy and safety of brexpiprazole for the treatment of adults experiencing an acute episode of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* The patient has schizophrenia, diagnosed according to DSM-IV-TR™ and confirmed by the Mini International Neuropsychiatric Interview (MINI).
* The patient has an acute exacerbation of psychotic symptoms and marked deterioration of usual function.
* The patient is willing to be hospitalised from the Screening Visit through Week 6.
* The patient will benefit from hospitalisation or continued hospitalisation for treatment of a current acute relapse of schizophrenia at study entry.
* The patient has a history of relapse and/or exacerbation of symptoms when not receiving antipsychotic treatment, excluding the current episode.
* The patient agrees to protocol-defined use of effective contraception.

Exclusion Criteria:

* The patient has a current Axis I diagnosis (DSM-IV-TR™ criteria) other than schizophrenia established as primary diagnosis.
* The patient suffers from a current Axis II diagnosis (DSM-IV-TR™ criteria).
* The patient suffers from mental retardation, organic mental disorders, or mental disorders due to a general medical condition (DSM-IV-TR™ criteria).
* The patient, in the opinion of the investigator or according to Columbia Suicide Severity Rating Scale (C-SSRS), is at significant risk of suicide.
* The patient has clinically significant tardive dyskinesia or severe akathisia at enrolment.
* The patient has a history of neuroleptic malignant syndrome.
* The patient has any relevant medical history or current presence of systemic disease.
* The patient has, at the Screening Visit an abnormal ECG or other abnormal ECG tests that are, in the investigator's opinion, clinically significant.
* The patient has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin, that has not been in remission for >5 years prior to the first dose of brexpiprazole.
* The patient is, in the investigator's opinion, unlikely to comply with the protocol or is unsuitable for any reason.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- US009, Escondido, California, United States

REFERENCES:
- [Derived] Ismail Z, Kapadia S, Palma AM, Yildirim M, Farovik A. Brexpiprazole for anxiety symptoms in schizophrenia: a pooled analysis of short- and long-term trials. Curr Med Res Opin. 2025 Aug;41(8):1535-1548. doi: 10.1080/03007995.2025.2552286. Epub 2025 Sep 11. PMID 40859756
- [Derived] Ismail Z, Meehan SR, Farovik A, Kapadia S, Palma AM, Zhang Z, McIntyre RS. Effects of brexpiprazole on patient life engagement in schizophrenia: post hoc analysis of Positive and Negative Syndrome Scale data. Curr Med Res Opin. 2025 Jan;41(1):145-153. doi: 10.1080/03007995.2024.2440059. Epub 2025 Jan 3. PMID 39749727
- [Derived] Correll CU, He Y, Therrien F, MacKenzie E, Meehan SR, Weiss C, Hefting N, Hobart M. Effects of Brexpiprazole on Functioning in Patients With Schizophrenia: Post Hoc Analysis of Short- and Long-Term Studies. J Clin Psychiatry. 2022 Mar 1;83(2):20m13793. doi: 10.4088/JCP.20m13793. PMID 35235720
- [Derived] Marder SR, Meehan SR, Weiss C, Chen D, Hobart M, Hefting N. Effects of Brexpiprazole Across Symptom Domains in Patients With Schizophrenia: Post Hoc Analysis of Short- and Long-Term Studies. Schizophr Bull Open. 2021 May 1;2(1):sgab014. doi: 10.1093/schizbullopen/sgab014. eCollection 2021 Jan. PMID 34901863
- See also: EMA EudraCT Results: 2012-002252-17 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2012-002252-17/results

RESULTS

PARTICIPANT FLOW:
Groups:
- Quetiapine Extended Release: Active Reference
  Quetiapine extended release: 400-800 mg/day, once daily, encapsulated tablets, orally
Period: Overall Study
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Started | 163 | 151 | 154
Treated | 161 | 150 | 153
Completed | 108 | 113 | 122
Not Completed | 55 | 38 | 32
Not completed — Randomised not treated | 2 | 1 | 1
Not completed — Adverse Event | 11 | 14 | 4
Not completed — Lack of Efficacy | 24 | 10 | 11
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 6 | 0 | 6
Not completed — Administrative or other reasons | 11 | 13 | 9

BASELINE CHARACTERISTICS:
Population: all-patients-treated set (APTS)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release | Total
Number analyzed (Participants) | 161 | 150 | 153 | 464
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.85 (10.56) | 39.68 (10.87) | 41.12 (10.91) | 40.56 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 66 | 64 | 200
  Male | 91 | 84 | 89 | 264
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 35 | 33 | 38 | 106
  White | 123 | 113 | 113 | 349
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 50 | 52 | 56 | 158
  Estonia | 4 | 3 | 4 | 11
  France | 1 | 0 | 1 | 2
  Poland | 5 | 5 | 5 | 15
  Romania | 14 | 13 | 11 | 38
  Serbia | 13 | 11 | 11 | 35
  Slovakia | 1 | 1 | 1 | 3
  Ukraine | 30 | 28 | 29 | 87
  Russian Federation | 43 | 37 | 35 | 115
Time since schizophrenia diagnosis (years) [Mean (Standard Deviation); unit: years] | 14.15 (9.35) | 12.88 (9.43) | 13.78 (9.49) | 13.62 (9.42)
Time since first antipsychotic treatment (years) [Mean (Standard Deviation); unit: years] | 14.48 (8.98) | 13.43 (9.19) | 14.31 (9.34) | 14.08 (9.16)
PANSS total score [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Syndrome Scale (PANSS) is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score (30 items) ranged from 30 to 210 with a higher score indicating greater severity of symptoms. PANSS total score is reported for the full analysis set (FAS); PBO=159, Brex=150, Que=150, and no total value was summarised for reporting
  units on a scale | 98.38 (10.30) | 97.82 (10.25) | 98.82 (10.83) | 98.34 (10.45)
CGI-S Score [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients). CGI-S score is reported for the full analysis set (FAS); PBO=159, Brex=150, Que=150, and no total value was summarised for reporting
  units on a scale | 4.94 (0.57) | 4.96 (0.59) | 4.98 (0.57) | 4.96 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in PANSS Total Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score (30 items) ranged from 30 to 210 with a higher score indicating greater severity of symptoms.
Time Frame: Baseline and Week 6
Population: Full-analysis set (FAS)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
units on a scale | -15.9 (1.5) | -20.0 (1.5) | -24.0 (1.5)
Statistical Analysis 1: Comparison: Placebo vs Brexpiprazole; The overall significance level was 0.05. The primary and the key secondary endpoints were tested hierarchically. Only if the primary endpoint was statistically significant would confirmatory testing continue with the key secondary endpoint; Test type: Superiority or Other; p = 0.0560, Mixed Models Analysis — For all efficacy analyses the primary comparison is the difference between brexpiprazole 2 to 4 mg/day and placebo at Week 6; Pooled site, visit, treatment as fixed effects, baseline score as continuous covariate, treatment-by-visit and baseline score-by-visit as interactions; Least square mean difference = -4.1, 95% CI 2-sided [-8.2 to 0.1], Standard Error of Mean 2.1
Statistical Analysis 2: Comparison: Placebo vs Quetiapine Extended Release; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Least square mean difference = -8.0, 95% CI 2-sided [-12.2 to -3.9], Standard Error of Mean 2.1

2. Secondary Outcome: Change From Baseline to Week 6 in CGI-S Score
Description: The Clinical Global Impression - Severity of Illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness.
  The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline and Week 6
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
units on a scale | -0.9 (0.1) | -1.2 (0.1) | -1.4 (0.1)

3. Secondary Outcome: CGI-I Score at Week 6
Description: The Clinical Global Impression - Global Improvement (CGI-I) provides the clinician's impression of the patient's improvement (or worsening).
  The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the rater believes the improvement is drug-related or not.
Time Frame: Week 6
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
units on a scale | 3.0 (0.1) | 2.7 (0.1) | 2.5 (0.1)

4. Secondary Outcome: Change From Baseline to Week 6 in PANSS Positive Subscale Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS Positive Subscale score is calculated from 7 items (for example: delusions, conceptual disorganization and hallucinatory behaviour). Symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. Higher score indicating greater severity of symptoms
Time Frame: Baseline and Week 6
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
units on a scale | -5.4 (0.5) | -7.0 (0.5) | -8.1 (0.5)

5. Secondary Outcome: Change From Baseline to Week 6 in PANSS Negative Subscale Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS Negative Subscale score is calculated from 7 items (for example: blunted affect, emotional withdrawal and poor rapport). Symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. Higher score indicating greater severity of symptoms
Time Frame: Baseline and Week 6
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
units on a scale | -3.1 (0.4) | -3.7 (0.4) | -4.5 (0.4)

6. Secondary Outcome: Change From Baseline to Week 6 in PANSS General Psychopathology Subscale Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS General Psychopathology Subscale score is calculated from 16 items (for example: somatic concern, anxiety and guilt feelings). Symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. Higher score indicating greater severity of symptoms
Time Frame: Baseline and Week 6
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
units on a scale | -8.2 (0.7) | -9.9 (0.7) | -11.6 (0.7)

7. Secondary Outcome: Change From Baseline to Week 6 in PANSS Excited Component Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS Excited Component score is calculated from 5 items (for example: poor impulse control, tension and hostility). Symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. Higher score indicating greater severity of symptoms
Time Frame: Baseline and Week 6
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
units on a scale | -2.5 (0.3) | -3.3 (0.3) | -3.9 (0.3)

8. Secondary Outcome: Change From Baseline to Week 6 in PANSS Marder Factor Scores: Negative Symptoms
Description: The Positive and Negative Syndrome Scale (PANSS) is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS Marder Factor scores: negative symptoms is calculated from 7 items (for example: blunted affect, emotional withdrawal and motor retardation). Symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. Higher score indicating greater severity of symptoms
Time Frame: Baseline and Week 6
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
units on a scale | -3.6 (0.4) | -4.3 (0.4) | -4.8 (0.4)

9. Secondary Outcome: Change From Baseline to Week 6 in PANSS Marder Factor Scores: Positive Symptoms
Description: The Positive and Negative Syndrome Scale (PANSS) is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS Marder Factor scores: positive symptoms is calculated from 8 items (for example: delusions, conceptual disorganization and stereotype thinking). Symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. Higher score indicating greater severity of symptoms
Time Frame: Baseline and Week 6
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
units on a scale | -5.7 (0.5) | -7.1 (0.5) | -8.4 (0.5)

10. Secondary Outcome: Change From Baseline to Week 6 in PANSS Marder Factor Scores: Disorganized Thoughts
Description: The Positive and Negative Syndrome Scale (PANSS) is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS Marder Factor scores: disorganized thoughts is calculated from 7 items (for example: conceptual disorganization, difficulty in abstract thinking and mannerisms and posturing). Symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. Higher score indicating greater severity of symptoms
Time Frame: Baseline and Week 6
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
units on a scale | -3.2 (0.4) | -4.0 (0.4) | -4.8 (0.3)

11. Secondary Outcome: Change From Baseline to Week 6 in PANSS Marder Factor Scores: Uncontrolled Hostility/Excitement
Description: The Positive and Negative Syndrome Scale (PANSS) is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS Marder Factor scores: uncontrolled hostility/excitement is calculated from 4 items (for example: excitement, hostility, and uncooperativeness).Symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. Higher score indicating greater severity of symptoms
Time Frame: Baseline and Week 6
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
units on a scale | -1.8 (0.3) | -2.5 (0.3) | -2.8 (0.3)

12. Secondary Outcome: Change From Baseline to Week 6 in PANSS Marder Factor Scores: Anxiety/Depression
Description: The Positive and Negative Syndrome Scale (PANSS) is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS Marder Factor scores: anxiety/depression is calculated from 4 items (for example: anxiety, guilt feelings, and tension). Symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. Higher score indicating greater severity of symptoms
Time Frame: Baseline and Week 6
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
units on a scale | -2.9 (0.2) | -3.2 (0.2) | -3.6 (0.2)

13. Secondary Outcome: Discontinuation Due to Lack of Efficacy During the Study
Description: Discontinuation due to lack of efficacy was based on the primary reason for withdrawal
Time Frame: Baseline to Week 6
Population: APTS
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 161 | 150 | 153
percentage of patients | 14.91 | 6.67 | 7.19

14. Secondary Outcome: Response Rate at Week 6
Description: The response rate was defined as a reduction of ≥30% from baseline in PANSS total score OR a CGI-I score of 1 or 2
Time Frame: Baseline and Week 6
Population: FAS (last assessment)
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 159 | 150 | 150
percentage of responders | 32.1 | 48.7 | 62.7

15. Secondary Outcome: Change From Baseline to Week 6 in PSP Total Score
Description: The Personal and Social Performance Scale (PSP) is a clinician-rated scale designed and validated to measure a patient's current level of social functioning. The PSP scale consists of a 100-point single-item rating scale, subdivided into 10 equal intervals. Scores of 1 to 10 indicate lack of autonomy in basic functioning, whereas scores of 91 to 100 reflect excellent functioning. The total score is rated by the investigator and is based on an algorithm which takes both the ratings of the 4 primary domains of PSP, and the combination of these ratings into account. The 4 primary domains are: socially useful activities (including work and study), personal and social relationships, self-care, and disturbing and aggressive behaviours. The 4 domains are assessed on a 6-point scale, from absent to very severe. A higher score indicates a better performance.
Time Frame: Baseline and Week 6
Population: FAS. PSP was collected at Baseline, Day 21 and Day 42 only, due to the windowing only patients with PSP assessments between Days 15 to 27 and after Day 35 were included in this analysis; the number of participants analysed is therefore smaller than the defined FAS and also smaller than other PSP analyses using LOCF.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 139 | 133 | 138
units on a scale | 9.4 (1.0) | 13.0 (1.0) | 15.3 (1.0)

16. Secondary Outcome: PSP Functional Remission Rate at Week 6
Description: The PSP functional remission rate was defined as a PSP total score ≥71
Time Frame: Week 6
Population: FAS (last assessment). Patients who have no post-baseline PSP values available were not included as response is defined based on change from baseline and no baseline carried forward analysis was planned; the number of participants analysed is therefore smaller than the defined FAS.
Measure: Number; unit: percentage of remitters
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 157 | 146 | 146
percentage of remitters | 5.7 | 9.6 | 14.4

17. Secondary Outcome: PSP Functional Response Rate at Week 6
Description: The PSP functional response rate was defined as ≥10 point improvement from Baseline on the PSP total score
Time Frame: Week 6
Population: as for outcome 16
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 157 | 146 | 146
percentage of responders | 36.3 | 53.4 | 64.4

18. Secondary Outcome: PSP Domain D: Disturbing and Aggressive Behaviours at Week 6
Description: PSP domain D: disturbing and aggressive behaviours were categorised as "aggressive" (corresponding to mild, manifest, marked, severe, or very severe) or "nonaggressive" (corresponding to absent)
Time Frame: Week 6
Population: FAS. As this was based on observed cases, only patients who have PSP assessment at Week 6 were included in this analysis; the number of participants analysed is therefore smaller than the defined FAS and also smaller than other PSP analyses where last assessment carried forward was used.
Measure: Number; unit: percentage of aggressive patients
Arm/Group | Placebo | Brexpiprazole | Quetiapine Extended Release
Number analyzed (Participants) | 112 | 114 | 126
percentage of aggressive patients | 30.4 | 27.2 | 22.2

ADVERSE EVENTS:
Time Frame: Baseline to end of treatment (Week 6)
Description: Treatment-Emergent Adverse Events are reported in this section
Groups:
- Quetiapine: Active Reference
  Quetiapine extended release: 400-800 mg/day, once daily, encapsulated tablets, orally
Arm/Group | Placebo | Brexpiprazole | Quetiapine
Serious Adverse Events (participants affected / at risk) | 6/161 | 7/150 | 2/153
Other Adverse Events (participants affected / at risk) | 44/161 | 48/150 | 73/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=161) | Brexpiprazole (N=150) | Quetiapine (N=153)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 1
Schizophrenia (Psychiatric disorders) | 4 | 3 | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=161) | Brexpiprazole (N=150) | Quetiapine (N=153)
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 13
Weight increased (Investigations) | 6 | 8 | 20
Akathisia (Nervous system disorders) | 4 | 9 | 6
Dizziness (Nervous system disorders) | 1 | 4 | 18
Headache (Nervous system disorders) | 11 | 8 | 9
Sedation (Nervous system disorders) | 5 | 4 | 8
Somnolence (Nervous system disorders) | 8 | 7 | 34
Insomnia (Psychiatric disorders) | 10 | 13 | 4
Schizophrenia (Psychiatric disorders) | 11 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No